CLINICAL TRIAL: NCT01742936
Title: Point of Care Testing for Coagulation Function Versus Standard Laboratory Testing in Pediatric Patients Undergoing Major Surgery
Brief Title: Point of Care Testing in Pediatric Patients Undergoing Major Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Vidya Raman, Director of Preoperative Assessment Testing, Nationwide Children's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB12-00762
Record Dates: First submitted 2012-12-03; First posted 2012-12-06 (Estimated); Results first posted 2016-06-08 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-07

CONDITIONS: Spinal Fusion; Cardiopulmonary Bypass
MeSH Terms: interventions — Laboratories, Hospital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spinal fusion (Experimental): Patients undergoing a posterior spinal fusion and having clotting factors checked by both hand held CoaguChek and Hospital Laboratory.
  Interventions: Device: CoaguChek; Other: Hospital Laboratory
- Cardiac bypass (Experimental): Patients undergoing surgery requiring cardiopulmonary bypass and having clotting factors checked by both hand held CoaguChek and Hospital Laboratory.
  Interventions: Device: CoaguChek; Other: Hospital Laboratory

INTERVENTIONS:
Device: CoaguChek — Hand held coagulation monitor.
Other: Hospital Laboratory — Coagulation testing done by hospital laboratory.

SUMMARY:
The current study proposes to investigate Point of Care Testing (POCT) (Coagcheck®) and compare obtained results versus standard laboratory coagulation parameters prothrombin time (PT) and partial thromboplastin time (PTT). The time difference in obtaining the two results will also be examined. A total of 100 pediatric patients undergoing spinal surgery or cardiopulmonary bypass will be enrolled and consented per protocol. Blood samples will be obtained simultaneously tested on both the standard laboratory apparatus and the Coagcheck® device. If the two results are comparable, this could have immediate clinical application and impact in the operating room as POCT results are available within 2-3 minutes compared to 1-2 hours for standard laboratory samples.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective posterior spinal fusion surgery at Nationwide Children's Hospital
* Parents willing & able to provide informed consent
* Child able to provide assent (if age appropriate)

Exclusion Criteria:

* Pre-existing bleeding disorders
* Any other circumstance which, in the opinion of the investigator, would put the patient at increased risk.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2013-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Spinal Fusion: Patients undergoing a posterior spinal fusion and having clotting factors checked by both hand held CoaguChek and Hospital Laboratory.
  CoaguChek
  Hospital Laboratory
Period: Overall Study
Arm/Group | Spinal Fusion | Cardiac Bypass
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spinal Fusion | Cardiac Bypass | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (2.2) | 9.4 (4.4) | 12 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 14 | 47
  Male | 17 | 36 | 53
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: International Normalized Ratio (INR) on CoaguChek
Description: Measuring the blood's ability to clot on a handheld monitor.
Time Frame: At end of surgery (an average of 2-4 hrs for cardiac bypass and 4-6 hrs. for spinal fusion)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Spinal Fusion | Cardiac Bypass
Number analyzed (Participants) | 49 | 38
ratio | 1.11 (0.07) | 4.6 (2.1)

2. Primary Outcome: International Normalized Ratio (INR) Performed by Hospital Laboratory
Description: Measuring the bloods ability to clot by the hospital's reference laboratory.
Time Frame: At end of surgery (an average of 2-4 hrs for cardiac bypass and 4-6 hrs. for spinal fusion)
Population: Three cases of device error with CoaguChek®, 1 insufficient blood for measurement in the laboratory, and 1 communication failure during sending the blood sample to the laboratory occurred leaving 87 patients for analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Spinal Fusion | Cardiac Bypass
Number analyzed (Participants) | 49 | 38
ratio | 1.2 (0.1) | 3.5 (3.2)

ADVERSE EVENTS:
Arm/Group | Spinal Fusion | Cardiac Bypass
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes